CLINICAL TRIAL: NCT03922932
Title: Wide-Field and Projection-Resolved Optical Coherence Tomography Angiography in Diabetic Retinopathy
Brief Title: WF and PR OCTA in Diabetic Retinopathy
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Thomas Hwang, MD, Associate Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: OHSU IRB#00016932
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; OCT; Angiography; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Group A: PDR: This group will consist of 30 subjects with active proliferative diabetic retinopathy (PDR) and 30 subjects with treated PDR.
- Group B: NPDR: This group will consist of 60 subjects with severe non-proliferative diabetic retinopathy (NPDR), 60 subjects with moderate NPDR, and 60 subjects with mild NPDR.
- Group ME: Macular Edema: This group is a sub-set of 25 subjects from either Group A or B who have macular edema requiring treatment.
- Group C: DM without Retinopathy: This group will consist of 60 subjects with diabetes mellitus (DM) who do not have retinopathy.
- Group D: Healthy Controls: This group will consist of 50 subjects with healthy eyes who do not have diabetes.

SUMMARY:
Diabetic retinopathy (DR) is a leading cause of vision loss in working-age Americans. Capillary damage from hyperglycemia causes vision loss through downstream effects, such as retinal ischemia, edema, and neovascularization (NV). Proper screening and timely treatment with laser photocoagulation and anti-vascular endothelial growth factor (VEGF) injections can minimize morbidity. In the last decade, clinicians have been able to use objective structural data from optical coherence tomography (OCT) to guide the treatment of diabetic macular edema. Other aspects of care, however, still largely depend on subjective interpretation of clinical features and fluorescein angiography (FA) to determine the disease severity and treatment threshold. The recently developed OCT angiography (OCTA) provides dye-less, injection-free, three-dimensional images of the retinal and choroidal circulation with high capillary contrast. Not only is it safer, faster, and less expensive than conventional dye-based angiography, OCTA provides the potential of giving clinicians objective tools for determining severity of disease by detecting and quantifying NV and non-perfusion.

ELIGIBILITY:
Participant-Related Inclusion Criteria:

I. All Diabetics (Groups A, B, C)

* Type 1 diabetes of at least 5 years duration or
* Type 2 diabetes of any duration II. Group B
* Able to return for follow-up over 3 years

Participant-Related Exclusion Criteria:

I. Group B

* Significant medical condition that would make long-term follow-up difficult II. Controls (Group D)
* Any medical problems associated with retinal vascular abnormalities (i.e., hypertension, systemic vasculitis, carotid insufficiency, etc.)

Eye-Related Inclusion Criteria:

I. Group A:

* Presence of active neovascularization, with or without prior treatment
* Presence of involuted fibrovascular proliferans

II. Group B:

* NPDR of any severity as defined by the International Clinical Diabetic Retinopathy Severity Scale

III. Groups C & D:

* No evidence of diabetic retinopathy

IV. Group ME:

* Presence of center-involving macular edema requiring treatment

Eye-Related Exclusion Criteria: (Applies to study eye only. May be present in non-study eye.)

* Visual acuity worse than 20/200
* Inability to maintain stable fixation for OCT imaging
* History of major eye surgery (vitrectomy, cataract surgery, scleral buckle, other intraocular surgery, etc.) within 90 days of enrollment
* History of another eye disease or condition that may alter retinal perfusion, permeability, or retinal anatomy
* Substantial media opacity (cataract, corneal scar, vitreous hemorrhage) that may interfere with study imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults age 18 or older with either healthy eyes or diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PR-OCTA Measure of Non-Perfusion Areas | 3 years
  Non-perfusion areas of the 3 retinal plexuses and choriocapillaris will be measured in mm2.
Non-PR-OCTA Measure of Retinal Non-Perfusion Areas | 1 year
  Non-perfusion areas of the 3 retinal plexuses will be measured in mm2.
Non-PR-OCTA Retinal Neovascularization Areas | 1 year
  Retinal neovascularization areas will be measured in mm2.
Structural OCT Cyst Volume | 1 year
  Cyst volume will be measured in mm3.
Structural OCT Retinal Thickening Area | 1 year
  The area of retinal thickening will be measured in mm2.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hwang, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States